CLINICAL TRIAL: NCT01448057
Title: A Prospective, Randomized, Investigator-Blind Study to Compare Three Days of Treatment With Paracetamol (500 mg) / Dimethindene Maleate (1 mg) / Phenylephrine Hydrochloride (10 mg) Tablets Versus Paracetamol 500 mg Alone in the Treatment of Nasal Congestion and Other Symptoms Due to Cold and Flu
Brief Title: Evaluation of Efficacy and Safety of Tablets of Paracetamol, Dimethindene Maleate and Phenylephrine Hydrochloride in Reducing Symptoms of Common Cold and Flu
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 381-A-301
Record Dates: First submitted 2011-10-05; First posted 2011-10-07 (Estimated); Results first posted 2017-01-13 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-01

CONDITIONS: Upper Respiratory Tract Infection; Nasal Congestion; Rhinorrhea; Sneezing
Keywords: Paracetamol; dimethindene maleate; phenylephrine hydrochloride; cold and flu symptoms
MeSH Terms: conditions — Respiratory Tract Infections; Nasal Obstruction; Rhinorrhea; Sneezing; Common Cold | interventions — Acetaminophen; Dimethindene; Phenylephrine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combination Product (Experimental): Paracetamol (500 mg)/dimethindene maleate (1 mg)/ phenylephrine hydrochloride (10 mg) tablets
  Interventions: Drug: Paracetamol (500 mg)/dimethindene maleate (1 mg)/ phenylephrine hydrochloride (10 mg) tablets
- Paracetamol tablets (Active Comparator): Paracetamol (500 mg) tablets
  Interventions: Drug: Paracetamol (500 mg) tablets

INTERVENTIONS:
Drug: Paracetamol (500 mg)/dimethindene maleate (1 mg)/ phenylephrine hydrochloride (10 mg) tablets — Paracetamol (500 mg)/dimethindene maleate (1 mg)/ phenylephrine hydrochloride (10 mg) tablets
  Arms: Combination Product
Drug: Paracetamol (500 mg) tablets — Paracetamol (500 mg) tablets
  Arms: Paracetamol tablets

SUMMARY:
The study is a clinical evaluation of an over the counter (OTC) combination product containing paracetamol (500 mg), dimethindene maleate (1 mg), phenylephrine hydrochloride (10 mg) compared to paracetamol (500 mg) alone in the treatment of nasal congestion, rhinorrhea, sneezing and other symptoms due to upper respiratory tract infection (URTI).

ELIGIBILITY:
* Inclusion criteria:

  • acute URTI, diagnosed by a health care professional at the study site, with the following symptoms having started within 72 hours before the screening/baseline Visit: nasal congestion, sneezing, and rhinorrhea.
* Exclusion criteria:

  * Use of other investigational drugs within 30 days or 10 half-lives before enrollment, whichever is longer.
  * History of or known hypersensitivity to any of the study drugs, excipients or to drugs of similar chemical classes.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 341 (Actual)
Dates: Start 2013-07; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- Brazil (6):
  - Santa Casa De Misericordia De Belo Horizonte - Avenida Francisco Sales 1111, Santa Efigenia, Belo Horizonte/MG
  - Sociedade Campineira De Educacao E Instrucao - Rodovia Dom Pedro I, KM 136 Parque das Universidades, Campinas/SP
  - Instituto de Ensino e Pesquisa Clínica do Ceará, Rua Coronel Jucá, 1952 - Dionísio Torres -, Fortaleza/CE
  - Polonio Clinica De Servicios Medicos EM Gastroenterologia E Cirurgia Toracica S/S LTDA - ME, Rua Major Alfredo Servulo de Oliveira Romao, 103, Chacara Braz Miraglia, Jau/SP
  - : Lal Clinica Centro de Pesquisa e Desenvolvimento Ltda, Rua General Osório, 503, Vila Martina / Valinhos, São Paulo
  - Associacao Fundo De Incentivo A Pesquisa - AFIP - Rua Marselhesa 500 - Vila Clementino, São Paulo

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Combination Product | Paracetamol Tablets
Started | 170 | 171
Completed | 162 | 167
Not Completed | 8 | 4
Not completed — Protocol Violation | 3 | 2
Not completed — Lost to Follow-up | 3 | 0
Not completed — Adverse Event | 0 | 2
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm A: Combination Product
  Paracetamol (500 mg)/dimethindene maleate (1 mg)/ phenylephrine hydrochloride (10 mg) tablets: Paracetamol (500 mg)/dimethindene maleate (1 mg)/ phenylephrine hydrochloride (10 mg) tablets
- Arm B: Paracetamol (500 mg) tablets
  Paracetamol (500 mg) tablets: Paracetamol (500 mg) tablets
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 170 | 171 | 341
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 170 | 171 | 341
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (11.64) | 34.5 (11.76) | 35.3 (11.71)
Gender [Count of Participants; unit: Participants]
  Female | 122 | 134 | 256
  Male | 48 | 37 | 85
Region of Enrollment [Number; unit: participants]
  Brazil | 170 | 171 | 341

OUTCOME MEASURES:

1. Primary Outcome: Physician Global Evaluation of Effectiveness on Nasal Symptoms
Description: The Physician will measure the reduction of Nasal Symptoms (Nasal Congestion, Sneezing, and Rhinorrhea) on day 2.
  Range from 1 to 5 where 1 is excellent and 5 is bad :
  1 = excellent : 75% to 100% remission of signs and symptoms 5 = bad : exacerbation of nasal symptoms
Time Frame: Day 2
Population: In the combination product arm 8 subjects had missing assessment and 1 subject in the paracetamol arm
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Arm A: Combination Product Paracetamol (500 mg)/dimethindene maleate (1 mg)/ phenylephrine hydrochloride (10 mg) tablets
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 162 | 170
score on a scale | 1.9 (0.84) | 2.1 (0.91)

2. Secondary Outcome: Daily Average of the Sum of a 100 mm Visual Analog Scale for All Symptoms
Description: Subject will assess Nasal and non Nasal symptoms using a 100 mm Visual Analog Scale for each symptom, 0=no symptoms 100= the worst possible symptoms
Time Frame: Day 3
Population: In the combination product arm 11 subjects had missing assessment and 5 subject in the paracetamol arm
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 159 | 166
mm | 169.2 (231.14) | 225.3 (262.59)

ADVERSE EVENTS:
Time Frame: 3 days
Arm/Group | Arm A | Arm B
Serious Adverse Events (participants affected / at risk) | 0/170 | 0/171
Other Adverse Events (participants affected / at risk) | 77/170 | 39/171
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=170) | Arm B (N=171)
somnolence (Nervous system disorders) | 71 (71) | 37 (37)
Abdominal pain (Gastrointestinal disorders) | 6 (6) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Preliminary agreement between Novartis Consumer Health and the investigator